CLINICAL TRIAL: NCT05193773
Title: The Effects of a Multifactorial Intervention to Reduce Physical Restraints for Care Providers in Nursing Homes: A Cluster Randomized Controlled Trial
Brief Title: Effects of a Multifactorial Intervention to Reduce Physical Restraints for Care Providers in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Su-Hua Liang (Other)
Responsible Party: Sponsor-Investigator, Su-Hua Liang, Investigator, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 104-5256B
Record Dates: First submitted 2022-01-05; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Nursing Homes; Intervention; Older People
Keywords: care providers; restraints

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comparison group (No Intervention): The Control Group received no extra care.
- Intervention Group (Experimental): Intervention Group, Intervention with follow-up, will have a multifactorial interventions to reduce physical restraint.
  Interventions: Other: multifactorial interventions

INTERVENTIONS:
Other: multifactorial interventions — The experimental group underwent multifactorial interventions to reduce physical restraint, including developing routines for physical restraint, promoting institutional policies to reduce the use of physical restraint, developing alternative methods, education, and consultations.
  Arms: Intervention Group

SUMMARY:
Scholars from around the world have been strongly advocating restraint-free care in long-term care institutions. Therefore, the aim of this study was to evaluate the effects of a multifactorial intervention to reduce physical restraints for care providers in nursing homes.

DETAILED DESCRIPTION:
In Taiwanese nursing homes, the use of physical restraints on residents as a protective measure is fairly common. However, physical restraints can be seen as a violation of human rights, and there is no guarantee of the effectiveness or safety of such physical restraints.This study was to evaluate the effects of a multifactorial intervention to reduce physical restraints for care providers in nursing homes. A cluster randomized controlled trial was conducted using pretest-posttest control group design. A purposive sampling of participants was chosen from care providers of 6 nursing home institutions in Taiwan, who were then randomly assigned to the experimental group (3 nursing homes) or the control group (3 nursing homes). The experimental group underwent multifactorial interventions to reduce physical restraint.

ELIGIBILITY:
Inclusion Criteria:

* A full-time care provider
* Worked in a nursing home for more than three months
* Care providers have imposed physical restraints on elderly residents aged 60 or above Within the last month.

Exclusion Criteria:

• can't speak or read chinese, Vietnamese, Indonesian

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
knowledge | 8 minutes
  The Knowledge of Restraints use scale . The Knowledge of Restraints use scale was used to assess the knowledge component. The scale consists of 20 items scored as 1 (true) or 0 (false or uncertainty). A higher score indicates more knowledge; total scores range from 0 to 20.
Attitudes | 8 minutes
  The Attitudes of Restraints use scale . The Attitudes of Restraints use scale was used to assess participants' attitudes about restraint use. The scale is a 15 items with a 5-point Likert scale ranging from 1 (not at all agree) to 5 (most agree); the range of total scores is from 15 to 75. Higher scores indicate more negative attitudes about physical restraint use.
Behavior | 4 minutes
  The Behavior of restraints use scale . The Behavior of restraints use scale was used to assess care providers' behavior about restraint use. The scale consists of 13 items scored as 1 (yes) or 0 (no); the range of total scores is from 0 to 13. The higher the score, the better the behavior.
physical restraint use | 1 minutes
  the percentage of physical restraint use

SECONDARY OUTCOMES:
Restraint types | 1 minutes
  The percentage of restraint types use. The restraint types including device (wrist belt, waist belt, ankle belt, vest in wheel chair, belt in wheel chair, wheel chair with a table board, hand mitts, special sheet etc), area (trunk, waist, ankle, wrist), belt in bed, belt in wheel chair, day time, night, whole day.
Multiple restraints | 1 minutes
  the percentage of multiple restraints
agitated and inappropriate behavior | 1 minutes
  the percentage of agitated and inappropriate behavior
Extubation rate | 1 minutes
  the percentage of extubation
falls rate | 1 minutes
  the percentage of falls
psychotropic medication prescriptions | 1 minutes
  the percentage of psychotropic medication prescriptions
fall-related fractures | 1 minutes
  the percentage of fall-related fractures

CONTACTS AND LOCATIONS:
Overall Officials: Su-Hua Liang, Principal Investigator
Locations (1):
- Nursing Homes, Miaoli, Taiwan